CLINICAL TRIAL: NCT02663297
Title: Phase I Study of the Administration of T Lymphocytes Expressing the CD30 Chimeric Antigen Receptor (CAR) for Prevention of Relapse of CD30+ Lymphomas After High Dose Therapy and Autologous Stem Transplantation (ATLAS)
Brief Title: Administration of T Lymphocytes for Prevention of Relapse of Lymphomas
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LCCC 1524-ATL; R01HL114564 (NIH)
Record Dates: First submitted 2016-01-17; First posted 2016-01-26 (Estimated); Results first posted 2025-05-15 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Hodgkin Disease; Lymphoma; Lymphoma, Non-Hodgkin; Immune System Diseases; Immunoproliferative Disorders; Lymphatic Diseases; Lymphoproliferative Disorders; Neoplasms; Neoplasms by Histologic Type
Keywords: CAR T cells; CD30; Lymphoma; T Lymphocytes
MeSH Terms: conditions — Hodgkin Disease; Lymphoma; Lymphoma, Non-Hodgkin; Immune System Diseases; Immunoproliferative Disorders; Lymphatic Diseases; Lymphoproliferative Disorders; Neoplasms; Neoplasms by Histologic Type

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ATLCAR.CD30 cells (Experimental): Three dose levels of ATLCAR.CD30 cells will be evaluated. Using the modified continual reassessment method (CRM), initial cohort of size two will be enrolled at each dose level after that subjects are enrolled one at a time until a minimum of 12 patients is treated. Each patient will receive one injection according to the dosing schedules listed below. Investigators will start with the lowest cell dose (2X10^7 cells/m^2) given to patients in one of our previous trials employing CAR-T cells including the CD28 costimulatory endodomain, and investigators will escalate the cell dose to the highest cell dose (2X10^8/m^2) given in the same trial.
  Note: Initially, only adults will be enrolled during the dose escalation phase of the study. Once a dose level has been tested in at least 2 adults without the occurrence of dose limiting toxicities (DLTs), children may then be enrolled on that dose level according to the CRM.
  Interventions: Drug: ATLCAR.CD30 cells

INTERVENTIONS:
Drug: ATLCAR.CD30 cells — Three dose levels will be evaluated:
  Group One, 2x10^7 cells/m^2 (maximum dose 5x10^7 cells)
  Group Two, 1x10^8 cells/m^2 (maximum dose 2.5x10^8 cells)
  Group Three, 2x10^8 cells/m^2 (maximum dose 5x10^8 cells)
  Other Names: CAR.CD30 T cells

SUMMARY:
The body has different ways of fighting infection and disease. No single way seems perfect for fighting cancer. This research study combines two different ways of fighting disease: antibodies and T cells. Antibodies are proteins that protect the body from disease caused by bacteria or toxic substances. Antibodies work by binding those bacteria or substances, which stops them from growing and causing bad effects. T cells, also called T lymphocytes, are special infection-fighting blood cells that can kill other cells, including tumor cells or cells that are infected. Both antibodies and T cells have been used to treat patients with cancers. They both have shown promise, but neither alone has been sufficient to cure most patients. This study is designed to combine both T cells and antibodies to create a more effective treatment. The treatment that is being researched is called autologous T lymphocyte chimeric antigen receptor cells targeted against the CD30 antigen (ATLCAR.CD30) administration.

In previous studies, it has been shown that a new gene can be put into T cells that will increase their ability to recognize and kill cancer cells. A gene is a unit of DNA. Genes make up the chemical structure carrying the patient's genetic information that may determine human characteristics (i.e., eye color, height and sex). The new gene that is put in the T cells in this study makes a piece of an antibody called anti-CD30. This antibody floats around in the blood and can detect and stick to cancer cells called lymphoma cells because they have a substance on the outside of the cells called CD30. Anti-CD30 antibodies have been used to treat people with lymphoma, but have not been strong enough to cure most patients. For this study, the anti-CD30 antibody has been changed so that instead of floating free in the blood part of it is now joined to the T cells. Only the part of the antibody that sticks to the lymphoma cells is attached to the T cells instead of the entire antibody. When an antibody is joined to a T cell in this way it is called a chimeric receptor. These CD30 chimeric (combination) receptor-activated T cells seem to kill some of the tumor, but they do not last very long in the body and so their chances of fighting the cancer are unknown.

The purpose of this research study is to determine a safe dose of the ATLCAR.CD30 cells that can be given to subjects after undergoing an autologous transplant. This is the first step in determining whether giving ATLCAR.CD30 cells to others with lymphoma in the future will help them. The researchers also want to find out what side effects patients will have after they receive the ATLCAR.CD30 cells post-transplant. This study will also look at other effects of ATLCAR.CD30 cells, including their effect on your cancer and how long they will survive in your body.

DETAILED DESCRIPTION:
STUDY OBJECTIVES

Primary Objective

* To determine the safety and tolerability and to estimate the MTD of ATLCAR.CD30 post ASCT in patients with CD30+ lymphoma at high risk for relapse

Secondary Objectives

* To measure the survival of ATLCAR.CD30 in vivo
* To estimate PFS after infusion of ATLCAR.CD30 post ASCT in patients with CD30+ lymphoma at high risk for relapse
* To determine the overall survival after infusion of ATLCAR.CD30 post ASCT in patients with CD30+ lymphoma at high risk for relapse

Exploratory Objective

* To measure patient-reported symptom, physical function, and health-related quality of life at baseline and over time in patients treated with ATLCAR.CD30 cells.

ENDPOINTS

Primary Endpoint

* Toxicity will be classified and graded according to the National Cancer Institute's Common Terminology Criteria for Adverse Events (CTCAE, version 4.0) and CRS toxicity will be graded according to the toxicity scale outlined in 11.6 (Appendix F: CRS Toxicity Grading Scale and Management Guidelines). The MTD will be based on the rate of dose-limiting toxicity

Secondary (Clinical) Endpoint

* PFS is defined from day of ASCT to relapse (in subjects with a documented complete response after ASCT) or progression (in subjects with documented stable disease or partial response after ASCT), or death as a result of any cause as per the Revised Response Criteria for Malignant Lymphoma.
* Overall survival will be measured from the date of administration of CAR.CD30 transduced ATL to date of death
* Persistence of CAR.CD30 T cells in vivo will be determined by quantitative PCR and flow cytometry in peripheral blood samples.

Exploratory Endpoint

* Patient reported symptoms will be measured using selected symptoms from the NCI PRO-CTCAE. Patient-reported physical function will be measured using the PROMIS Physical Function Score derived from the PROMIS Physical Function Short Form 20a v1.0. Patient-reported health-related quality of life will be measured using the PROMIS Global Health Score derived from the PROMIS Global Health Short Form v1.0-1.1.

OUTLINE

Patients scheduled to undergo an autologous stem cell transplantation (ASCT) for treatment of lymphoma will be approached for consent to screening and potential enrollment into LCCC1524. Peripheral blood cells will be collected from consenting patients who meet eligibility for cell procurement for creation of ATLCAR.CD30 cells prior to ASCT. The ASCT, including mobilization and collection of PBSCs, administration of myeloablative therapy, reinfusion of PBSCs and supportive care following transplant will be as per routine standard of care, and not expected to be impacted by enrollment into LCCC1524. Post ASCT, patients who meet eligibility criteria for treatment will receive one infusion of ATLCAR.CD30 cells once there is evidence of hematologic recovery. Research personnel will keep track of any patients who undergo procurement but do not undergo treatment with ATLCAR.CD30 cells, and the reason for withholding treatment.

Cell Procurement

Peripheral blood, up to 300 mL total (in up to 3 collections) will be obtained for subjects for cell procurement. In patients with low (CD3 count as assayed by flow cytometry less than 200/μl) T-cell count in the peripheral blood, a leukopheresis may be performed to isolate sufficient T cells. The parameters for pheresis will be up to 2 blood volumes.

For pediatric patients (patients under 18 years of age), the total amount of blood drawn will not be more than 3 mL (less than 1 teaspoon per 2.2 lbs. that the child weighs.

ATLCAR.CD30 Cells Administration

Post ASCT, once the patient has started to experience hematologic recovery (defined as ANC ≥500 cells/mm3 for 3 consecutive days, AND platelet count ≥25 cells/mm3 without transfusion over the preceding 5 days, AND Hg ≥8g/dL without transfusion support over preceding 5 days), ATLCAR.CD30 cells will be admnistered. This will generally occur between 14 and 20 days following infusion of autologous stem cells following high-dose chemotherapy.

Duration of Therapy

Therapy in LCCC1524 involves just one infusion of ATLCAR.CD30 cells. Treatment with one infusion will be administered unless:

* Patient decides to withdraw from study treatment, OR
* General or specific changes in the patient's condition render the patient unacceptable for further treatment in the judgment of the investigator.

Duration of Follow-Up

Patients will be followed for up to 15 years or until death, whichever occurs first. Patients removed from study for unacceptable adverse events will be followed until resolution or stabilization of the adverse event.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent explained to, understood by and signed by patient/guardian; patient/guardian given copy of informed consent.
* 3 to 17 years of age for pediatric patients, ≥18 years of age for adults; NOTE: children will not be allowed to enroll in a dose cohort until a minimum of 2 adult subjects are enrolled and complete their DLT assessment follow-up at that dose level
* Diagnosis of recurrent HL with a treatment plan that will include high dose chemotherapy with/without total body irradiation and autologous cell transplantation
* NHL patients with ALK negative CD30+ anaplastic large-cell lymphomas, CD30+ ALCL regardless of ALK status, with chemotherapy-sensitive relapse, CD30+ high-risk DLBCL, CD30+ cutaneous T cell lymphoma, or CD30+ mycosis fungoides who are otherwise eligible for transplant, are eligible for this study
* CD30+ disease (result can be pending at the time of cell procurement, but must be confirmed prior to treatment with ATLCAR.CD30 cells); NOTE: CD30 + disease is defined as requiring documentation of CD30 expression by immunohistochemistry based on the institutional hematopathology standard.
* Evidence of adequate organ function as defined by:

  * The following is required prior to procurement (NOTE: labs do not need to be redrawn if they have already been performed as part of SOC pre-transplant work-up; Subject must be eligible to receive ASCT)

    * Hgb ≥ 8.0g/dL
    * Bilirubin ≤1.5 times the upper limit of normal (ULN)
    * AST ≤ 3 times ULN
    * Serum creatinine ≤1.5 times ULN
    * Cardiac and pulmonary function that is adequate for ASCT
  * The following is required prior to infusion of ATLCAR.CD30 cells:

    * Absolute neutrophil count (ANC) ≥500 cells/mm^3 for 3 consecutive days; Note: ANC may be measured at the beginning and the end of a time frame expanding at least 3 days and does not need to be evaluated on each individual day AND
    * Platelet count ≥25,000 cells/mm^3 without transfusion over preceding 5 days Note: Platelets may be measured at the beginning and the end of a time frame expanding at least 5 days and does not need to be evaluated on each individual day AND
    * Hg ≥8g/dL without transfusion support over preceding 5 days Note: Hg may be measured at the beginning and the end of a time frame expanding at least 3 days and does not need to be evaluated on each individual day
    * Bilirubin ≤1.5 times the upper limit of normal (ULN)
    * AST ≤ 3 times ULN
    * Serum creatinine ≤1.5 times ULN
    * Pulse oximetry of > 90% on room air
* Imaging results from within 60 days prior to transplant (used as baseline measure for documentation of disease status). Note: Results may be obtained at a time point greater than 30 days from transplant if obtained per the patient's standard of care and with prior sponsor approval.
* Negative serum pregnancy test within 72 hours prior to procurement and again 72 hours prior to infusion
* Karnofsky or Lansky score of > 60%
* Considered at high risk for relapse as defined by: The presence of ≥ 1 of the following: failure to achieve CR post initial treatment; relapsed disease with an initial remission duration of <12 months; or extranodal involvement at the start of pre-transplant salvage therapy
* Subjects must have autologous transduced activated T cells that meet the Certificate of Analysis (CoA) acceptance criteria
* Women of childbearing potential (WOCBP) should be willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study, and for 6 months after the study is concluded. WOCBP are those who have not been surgically sterilized or have not been free from menses for > 1 year. The two birth control methods can be composed of: two barrier methods or a barrier method plus a hormonal method to prevent pregnancy. The male partner of WOCBP subjects enrolled into the trial should be instructed to use a condom by their female partner enrolled in the trial.

Exclusion Criteria:

* Received any investigational agents or received any tumor vaccines within the previous six weeks prior to cell infusion.
* Received anti-CD30 antibody-based therapy within the previous 4 weeks prior to cell infusion
* History of hypersensitivity reactions to murine protein-containing products
* Pregnant or lactating
* Tumor in a location where enlargement could cause airway obstruction.
* Current use of systemic corticosteroids at doses ≥10mg/day prednisone or its equivalent; those receiving <10mg/day may be enrolled at discretion of investigator
* Active infection with HIV, HTLV, HBV, HCV (can be pending at the time of cell procurement; only those samples confirming lack of active infection will be used to generate transduced cells) . Active infection is defined as not being well controlled on therapy (Note: To meet eligibility subjects are required to be negative for HIV antibody or HIV viral load, negative for HTLV1 and 2 antibody, negative for Hepatitis B surface antigen, or negative for HCV antibody or HCV viral load).

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2016-06-07 (Actual); Primary Completion 2021-01-15 (Actual); Study Completion 2037-01 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Natalie Grover, MD, Principal Investigator — Clinical Director of Cellular Therapy Program
Locations (2):
- United States (2):
  - Lineberger Comprehensive Cancer Center at University of North Carolina - Chapel Hill, Chapel Hill, North Carolina
  - Wake Forest University, Winston-Salem, North Carolina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Grover NS, Hucks G, Riches ML, Ivanova A, Moore DT, Shea TC, Seegars MB, Armistead PM, Kasow KA, Beaven AW, Dittus C, Coghill JM, Jamieson KJ, Vincent BG, Wood WA, Cheng C, Morrison JK, West J, Cavallo T, Dotti G, Serody JS, Savoldo B. Anti-CD30 CAR T cells as consolidation after autologous haematopoietic stem-cell transplantation in patients with high-risk CD30+ lymphoma: a phase 1 study. Lancet Haematol. 2024 May;11(5):e358-e367. doi: 10.1016/S2352-3026(24)00064-4. Epub 2024 Mar 28. PMID 38555923
- See also: UNC Lineberger Comprehensive Cancer Center — http://unclineberger.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between June 7, 2016, and Nov 30, 2020, 18 participants were enrolled.
Pre-assignment Details: 18 patients were found eligible and started the study in 2 centers in the United States.
Groups:
- Dose Level 1: Each patient will receive one injection of cell dose 2 × 10^7 CAR T cells per square meter.
- Dose Level 2: Each patient will receive one injection of cell dose 1 × 10^8 CAR T cells per square meter.
- Dose Level 3: Each patient will receive one injection of cell dose 2 × 10^8 CAR T cells per square meter.
Period: Overall Study
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level 3
Started | 4 | 5 | 9
Completed | 4 | 5 | 9
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Participants who started to study treatment.
Groups:
- Level 1: Each patient will receive one injection of cell dose 2 × 10^7 CAR T cells per square meter.
- Level 2: Each patient will receive one injection of cell dose 1 × 10^8 CAR T cells per square meter.
- Level 3: Each patient will receive one injection of cell dose 2 × 10^8 CAR T cells per square meter.
- Total: Total of all reporting groups
Arm/Group | Level 1 | Level 2 | Level 3 | Total
Number analyzed (Participants) | 4 | 5 | 9 | 18
Age, Continuous [Mean (Full Range); unit: years] | 29.04 [20 to 49] | 35.12 [17 to 74] | 50.30 [17 to 77] | 41.34 [17 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 2 | 3
  Male | 3 | 5 | 7 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 4 | 5 | 9 | 18
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 1
  White | 3 | 5 | 7 | 15
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 4 | 5 | 9 | 18

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events as a Measure of Safety and Tolerability of Escalating Doses of Autologous Activated T Lymphocytes
Description: The Maximum tolerated dose was based on the rate of dose-limiting toxicity. Toxicity was classified and graded according to the National Cancer Institute's Common Terminology Criteria for Adverse Events (CTCAE, version 4.0), and cytokine release syndrome (CRS). The number of subjects with dose-limiting toxicity was recorded.CTCAE Grade 1 Mild, Grade 2 Moderate, Grade 3, Grade 4 Life-threatening consequences; urgent intervention indicated. Grade 5 Death related to AE. Cytokine Release Syndrome (CRS) will be graded according to American Society for Transplantation and Cellular Therapy (ASTCT) CRS Consensus Grading. Grade 1 - Mild Grade 2 - Moderate, Grade 3 - Severe (Aggressive Intervention): Grade 4 - Life-threatening (Life-sustaining intervention): Fever ≥38oC, Hypotension requiring multiple vasopressors, Hypoxia requiring positive pressure (e.g., CPAP, BiPAP, intubation, mechanical ventilation), Grade 5 - Death: Death.
Time Frame: 6 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Level 1 | Level 2 | Level 3
Number analyzed (Participants) | 4 | 5 | 9
Participants | 0 | 0 | 0

2. Secondary Outcome: To Measure the Survival of ATLCAR.CD30 in Vivo
Description: Persistence of CAR.CD30 T cells in vivo will be determined by quantitative polymerase chain reaction (PCR) and flow cytometry in peripheral blood samples
Time Frame: 15 years
Reporting Status: Not Posted

3. Secondary Outcome: To Estimate PFS After Infusion of ATLCAR.CD30 Post ASCT in Patients With CD30+ Lymphoma at High Risk for Relapse
Description: PFS is defined from day of ASCT to relapse (in subjects with a documented complete response after ASCT) or progression (in subjects with documented stable disease or partial response after ASCT), or death as a result of any cause as per the Revised Response Criteria for Malignant Lymphoma
Time Frame: 15 years
Reporting Status: Not Posted

4. Secondary Outcome: Determine the Overall Survival After Infusion of ATLCAR.CD30
Description: Overall survival will be measured from the date of administration of CAR.CD30 transduced ATL to date of death
Time Frame: 15 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse events were collected from day one of the study drug administration to 30 days after completion of treatment. (Up to 3 years)
Description: National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE v4.03).
Arm/Group | Level 1 | Level 2 | Level 3
All-Cause Mortality (participants affected / at risk) | 1/4 | 1/5 | 2/9
Serious Adverse Events (participants affected / at risk) | 0/4 | 1/5 | 0/9
Other Adverse Events (participants affected / at risk) | 4/4 | 5/5 | 9/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Level 1 (N=4) | Level 2 (N=5) | Level 3 (N=9)
Fever (General disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Level 1 (N=4) | Level 2 (N=5) | Level 3 (N=9)
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 2 | 1 | 0
Anemia (Blood and lymphatic system disorders) | 2 | 2 | 3
Anorexia (Metabolism and nutrition disorders) | 0 | 2 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 3 | 2 | 2
Blood bilirubin increased (Investigations) | 0 | 0 | 1
Blurred vision (Eye disorders) | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Creatinine increased (Investigations) | 0 | 1 | 0
Diarrhea (Gastrointestinal disorders) | 1 | 2 | 3
Dizziness (Nervous system disorders) | 1 | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Fatigue (General disorders) | 0 | 3 | 4
Fever (General disorders) | 0 | 0 | 1
Flu like symptoms (General disorders) | 0 | 0 | 1
General disorders and administration site conditions - Other, specify (General disorders) | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 1 | 2
Hypermagnesemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypernatremia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 | 1 | 1
Hypocalcemia (Metabolism and nutrition disorders) | 0 | 1 | 3
Hypokalemia (Metabolism and nutrition disorders) | 0 | 1 | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 0 | 2 | 1
Hyponatremia (Metabolism and nutrition disorders) | 1 | 1 | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 0 | 1
Investigations - Other, specify (Investigations) | 0 | 1 | 1
Lymphocyte count decreased (Investigations) | 3 | 3 | 9
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2
Nausea (Gastrointestinal disorders) | 2 | 2 | 4
Neuralgia (Nervous system disorders) | 0 | 1 | 0
Neutrophil count decreased (Investigations) | 2 | 2 | 4
Neutrophil count decreased (Investigations) | 2 | 2 | 6
Non-cardiac chest pain (General disorders) | 0 | 1 | 0
Platelet count decreased (Investigations) | 2 | 4 | 5
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 2
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Treatment related secondary malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2
Tremor (Nervous system disorders) | 1 | 0 | 1
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 2 | 1
Weight loss (Investigations) | 0 | 1 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
White blood cell decreased (Investigations) | 2 | 3 | 7
hypotension (Vascular disorders) | 0 | 2 | 1
confusion (Psychiatric disorders) | 0 | 1 | 0
oral pain (Gastrointestinal disorders) | 0 | 0 | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Cytokine release syndrome (Immune system disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Subcontractor agrees that the first publication of the Study results will be made by Institution as a multi-site publication. Subcontractor can publish its site-specific results after Institution's publication, 12 months post-study completion, or upon Institution's notice of completion. Subcontractor must provide Institution 30 days for manuscript review and may delay publication for 45 days for institution's patent filing. Institution will register the Study and post results as required by law.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-04-17): https://cdn.clinicaltrials.gov/large-docs/97/NCT02663297/Prot_SAP_000.pdf